CLINICAL TRIAL: NCT02004600
Title: Bicentric, Open and Pilot Study Evaluating the Efficiency and the Tolerance of the Photodynamic Therapy in the Treatment of Epidermal Dysplasia for Patients Affected by Hereditary Dystrophic Epidermolysis Bullosa
Brief Title: Pilot Study Evaluating the Efficiency and the Tolerance of the PDT in the Treatment of Epidermal Dysplasia for Patients Affected by Hereditary DEB
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: health statement of pre-screenined patients were too bad for being enrolled in the study
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-AOI-11
Record Dates: First submitted 2013-11-26; First posted 2013-12-09 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Dystrophic Epidermolysis Bullosa
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica | interventions — Photochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- patient receiving one PDT session (Experimental): patient receiving one photodynamic therapy (PDT) session
  Interventions: Procedure: Photodynamic therapy (PDT)

INTERVENTIONS:
Procedure: Photodynamic therapy (PDT) — 1 session of Photodynamic therapy (PDT) on epidermis dysplasia
  Other Names: 1 session of Photodynamic therapy (PDT)

SUMMARY:
The hereditary dystrophic epidermolysis bullosa are genodermatosis responsible of a poor adhesion of the epidermis to the dermis pulling a large mucocutaneous fragility and recurrent spontaneous or posttraumatic bullous detachment. They are caused by mutations in the COL7A1 gene encoding for the collagen VII.

No curative treatment is avaible. The main cause of patients death is the development of squamous cell carcinoma, sometimes multiple and paticularly aggressive in repeated healing part. The photodynamic therapy (PDT) is one of technical reference of multiple actinic keratoses lesions for adults, which are also pre-epithelioma lesions. The PDT is well tolerated even by the elderly and requires only a single session.

The main objective of this study is to determine the efficiency of the photodynamic therapy in the treatment of epidermic dysplasies for patients affected by dystrophic epidermolysis bullosa (DEB). The secondary objectives are to evaluate the tolerance of this treatment in terms of pain and healing, and to evaluate the contribution of confocal microscopy in the diagnosis of epidermal dysplasia for patients affected by hereditary dystrophic epidermolysis bullosa. The main evaluation criterion is the cutaneous biopsy before and after (M2) a PDT session of an epidermal dysplasia area. The secondary criteria are the evaluation of the pain during the PDT session and the healing of the cutaneous lesion at M0, M2 and M4 (lesion area and healing time) and correlation histology / MC. Each patient with a suspicious lesion will be biopsied. In case of agreement for this protocol, there will be 1 PDT session followed by a consultation of control at 2 and 4 months after the end of treatment.

DETAILED DESCRIPTION:
The hereditary dystrophic epidermolysis bullosa are genodermatosis responsible of a poor adhesion of the epidermis to the dermis pulling a large mucocutaneous fragility and recurrent spontaneous or posttraumatic bullous detachment. They are caused by mutations in the COL7A1 gene encoding for the collagen VII.

No curative treatment is avaible. The main cause of patients death is the development of squamous cell carcinoma, sometimes multiple and paticularly aggressive in repeated healing part. The early treatment of pre-epithelioma cutaneous lesions to moderate at severe dysplasia type would undoubtedly allow to improve the prognosis of patients. Because of the cutaneous fragility of patients, topical treatments such as imiquimod or 5-FU are not possible. The photodynamic therapy (PDT) is one of technical reference of multiple actinic keratoses lesions for adults, which are also pre-epithelioma lesions. The PDT is well tolerated even by the elderly and requires only a single session.

The main objective of this study is to determine the efficiency of the photodynamic therapy in the treatment of epidermic dysplasies for patients affected by dystrophic epidermolysis bullosa (DEB). The secondary objectives are to evaluate the tolerance of this treatment in terms of pain and healing, and to evaluate the contribution of confocal microscopy in the diagnosis of epidermal dysplasia for patients affected by hereditary dystrophic epidermolysis bullosa. The main evaluation criterion is the cutaneous biopsy before and after (M2) a PDT session of an epidermal dysplasia area. The secondary criteria are the evaluation of the pain during the PDT session and the healing of the cutaneous lesion at M0, M2 and M4 (lesion area and healing time) and correlation histology / MC. This is a bicentric, open and pilot study on 5 patients over 18 years affected by hereditary dystrophic epidermolysis bullosa with epidermal displasia. Carcinomas in situ were excluded of this study. Each patient with a suspicious lesion will be biopsied. In case of agreement for this protocol, there will be 1 PDT session followed by a consultation of control at 2 and 4 months after the end of treatment.

Total study duration: 18 months (12 months for inclusions, 4 months for study, 2 months for data analysis).

ELIGIBILITY:
Inclusion Criteria:

* Patient carrying a widespread EBDR with moderate to severe epidermal dysplasia on a cutaneous biopsy of a suspicious lesion. Any clinically suspicious lesion should be biopsied in these patients, the inclusion will be made only after obtaining the results of the histological examination.
* The size of the lesion will be between 10 cm² and 1cm².
* Systematic Obtaining of the signed informed consent
* Patient affiliated to Social Security

Exclusion Criteria:

* Pregnant or lactating women.
* Patients unable to cooperate for all the duration of the study.
* Squamous cell carcinoma in situ or invasive on biopsy.
* Patient treated by chemotherapy for another reason.
* Contraindication at the PDT, patient unable to lie over an hour.
* Contraindication at fentanyl ( 50mcg Instanyl ) intra nasal :

oHypersensitivity to the active substance or to any of the excipients oUse in patients who have never received opioid treatment. oSevere respiratory depression or severe airway obstruction. oPrevious radiotherapy of the face. oRecurrent episodes of epistaxis oConcomitant administration of monoamine oxidase inhibitors, of potent CYP 3A4 inhibitors, of nasal decongestants, or other drugs (other than oxymetazoline ) administered by nasal way.

oSevere hepatic or renal insufficiency.

•Patients who have participated in a clinical trial in the previous 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-12; Primary Completion 2014-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Histological examination of a cutaneous biopsy | 2 MONTHS AFTER ENROLLMENT
  Histological examination of a cutaneous biopsy at M2 on the epidermal dysplasia area treated with PDT session

SECONDARY OUTCOMES:
Tolerance of PDT | every 10 minutes during PDT session
  Tolerance of PDT : evaluation of pain every 10 minutes during PDT session

CONTACTS AND LOCATIONS:
Overall Officials: Christine CHIAVERINI, MD, Principal Investigator — Nice University Hospital
Locations (2):
- France (2):
  - Nice University Hospital, Nice
  - Saint Louis Hospital, Paris